CLINICAL TRIAL: NCT04206865
Title: Prospective Comparison of ARNI to Alternate Oral Vasodilator Therapies to Determine the Hemodynamic Profile and Relative Tolerability of (ARNIs) in Patients With Decompensated Heart Failure and Low Cardiac Output
Brief Title: Comparison of ARNI to Alternate Oral Vasodilator Therapies in Patients With Low Cardiac Output
Acronym: PARAVLO-HF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: New study initiated
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Randall C Starling MD MPH, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1133
Record Dates: First submitted 2019-12-11; First posted 2019-12-20 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Cardiogenic Shock
Keywords: ARNI; Sacubitril-Valsartan; Cardiogenic Shock; Tailored Therapy; Cardiac Intensive Care
MeSH Terms: conditions — Shock, Cardiogenic | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARNI therapy (Experimental): Patient's randomized to this arm will receive sacubitril-valsartan per study protocol and titrated per titration guidelines.
  Interventions: Drug: Sacubitril-Valsartan
- Standard Oral Vasodilator (Active Comparator): Patient's randomized to this arm will receive the oral vasodilator that the clinician chooses including angiotensin receptor blocker (ARB), isosorbide dinitrate, hydralazine, and angiotensin-converting enzyme inhibitor (ACEi).
  Interventions: Drug: Standard Oral Vasodilators

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Patient's will be randomized to ICU initiation of sacubitril-valsartan vs. alternate oral vasodilator therapy in 1:1 fashion
  Other Names: ARNI therapy
  Arms: ARNI therapy
Drug: Standard Oral Vasodilators — Patient's will be randomized to ICU initiation of sacubitril-valsartan vs. alternate oral vasodilator therapy in 1:1 fashion. Alternate vasodilators will include ARBs, hydralazine and isosorbide dinitrate, and ACEi
  Other Names: Usual Care
  Arms: Standard Oral Vasodilator

SUMMARY:
This is a prospective, randomized, non-blinded, single-center efficacy study of acutely decompensated heart failure patients with reduced ejection fraction (HFrEF), low cardiac index (<2.2) as determined by pulmonary artery catheter (PAC) who have been hemodynamically stabilized and ready for transition to oral vasodilator therapy at the discretion of the clinician. The investigators would like to accomplish the following objectives with this study:

1. Establish the superiority of an upfront initiation strategy for sacubitril-valsartan at maintaining patients on ARNI therapy at one-month follow-up compared to usual care.
2. Establish the safety of initiating sacubitril-valsartan in an intensive care setting
3. Characterize the hemodynamic effect of sacubitril-valsartan on patients with low cardiac output
4. Expand the population of hospitalized patients that can be initiated on ARNIs and thus facilitate prior to hospital discharge patients who are on optimal goal-directed medical therapy (GDMT) for heart failure

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded, single-center efficacy study of acutely decompensated heart failure patients with reduced ejection fraction (HFrEF), low cardiac index (<2.2) as determined by pulmonary artery catheter (PAC) who have been hemodynamically stabilized and ready for transition to oral vasodilator therapy at the discretion of the clinician. The investigators would like to accomplish the following objectives with this study:

1. Establish the superiority of an upfront initiation strategy for sacubitril-valsartan at maintaining patients on ARNI therapy at one-month follow-up compared to usual care.
2. Establish the safety of initiating sacubitril-valsartan in an intensive care setting
3. Characterize the hemodynamic effect of sacubitril-valsartan on patients with low cardiac output
4. Expand the population of hospitalized patients that can be initiated on ARNIs and thus facilitate prior to hospital discharge patients who are on optimal goal-directed medical therapy (GDMT) for heart failure

In this pragmatic study, the primary endpoint will be establishing the superiority of sacubitril-valsartan as an oral vasodilator in maintaining ARNI therapy at one-month post hospital discharge as compared to usual care. Given the overall mortality and heart failure hospitalization benefit of ARNI over ACEI and other vasodilators has been established in large-scale clinical trials, establishing that upfront initiation of ARNI therapy in patients with low cardiac output is safe and can be maintained post-discharge would be of significant clinical benefit. Adverse events including symptomatic hypotension (requiring cessation of drug), development of worsening renal function (requiring cessation of drug), hyperkalemia [moderate (> 5.5 mmol/L) or severe (> 6 mmol/L)], or re-initiation of IV vasodilator or IV inotropic therapy will be monitored and tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Heart Failure with reduced ejection fraction (EF <40%) documented in past 1 year
2. Presence of low cardiac index ≤2.2 based on PA catheter measurement followed by stabilization and readiness to transition to oral vasodilator therapy
3. SBP > 90 and SVR >950 at the time of randomization or tolerating an adequate amount of IV vasodilator therapy i.e. sodium nitroprusside (clinician discretion) without symptomatic or sustained hypotension (>30 minutes)
4. Intention to maintain pulmonary artery catheter for hemodynamic directed optimization of therapy

Exclusion Criteria:

1. Acute kidney injury (increase in serum creatinine concentration of >0.5 mg per deciliter) and a decrease in the estimated GFR >25% in the preceding 24 hours
2. Documented intolerance to sacubitril, valsartan, or any ARBs, neprilysin inhibitors or any of the sacubitril/valsartan excipients, any history of angioedema
3. End-stage renal disease at screening, or estimated GFR <30mL/min/1.73m² by MDRD
4. Sustained Symptomatic hypotension after initiation of nitroprusside (Clinician Discretion or >30 minutes)
5. Acute Coronary Syndrome, Stoke, TIA, Cardiac, Carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within 3 months of screening
6. Hyperkalemia- Serum Potassium >5.5 mmol/L at randomization
7. Enrollment in concurrent clinical trials with investigational drugs
8. CAD likely to require surgical or percutaneous intervention within 3 months after screening
9. Implantation ofCRT, or upgrade of existing device or revision of the device leads within 1 month of screening
10. Heart Transplant or VAD or intent to transplant (on transplant list) or implant VAD in the next 6 months.
11. PI discretion regarding eligibility
12. Active infection/sepsis
13. Active use of temporary mechanical support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on ARNI therapy at one-month follow-up | 1 month
  This will be the proportion of patients randomized to each arm who remain on ARNI therapy at one-month follow-up. Reasons for discontinuation will be tracked.

SECONDARY OUTCOMES:
Length of time of in the Intensive Care Unit | Hospital discharge, 1 Month
  Length of time from admission to the cardiac intensive care unit to disposition.
Length of Hospital Stay | Hospital discharge, 1 Month
  Length of time in days from hospital admission to discharge.
Change in NT-proBNP from admission at one-month follow-up | 1 Month
  NT-proBNP value on admission and again drawn at the one-month follow-up visit.
30 day HF readmissions | 1 Month
  This includes 24 hr admits, IV therapy, ER visits for HF treatment that occur within 30 days of hospital discharge.
180 day telephone follow up to determine: ARNI yes or no, hospitalizations, mortality, LVAD or transplant | 180 days
  180 day telephone follow up to determine: ARNI yes or no, hospitalizations, mortality, LVAD or transplant

CONTACTS AND LOCATIONS:
Overall Officials: Randall Starling, MD, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States